CLINICAL TRIAL: NCT01611545
Title: Can Pharmacogenomic Testing Improve Response and Avoid Adverse Effects With Clopidogrel Therapy? A Biospecimen Bank for Genetic and Genomic Investigation of Clopidogrel.
Brief Title: Pharmacogenomics and Effective Treatment With Clopidogrel
Status: Completed | Type: Observational
Sponsor: Avera McKennan Hospital & University Health Center (Other)
Collaborators: Avera Heart Hospital of South Dakota (Unknown); North Central Heart Institute (Unknown)
Responsible Party: Sponsor
Other Study IDs: AIHG-1410-Clopidogrel
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Pharmacogenomics and Cardiovascular Events
Keywords: Pharmacogenomics; Pharmacogenetics; Clopidogrel; Plavix
MeSH Terms: interventions — Pharmacogenomic Testing; Clopidogrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood or buccal samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Clopidogrel: Patients taking or prescribed clopidogrel or under consideration Utilizing pharmacogenomics to determine the most effective treatment
  Interventions: Genetic: Pharmacogenomics

INTERVENTIONS:
Genetic: Pharmacogenomics — Utilizing pharmacogenomics to determine the most effective treatment
  Other Names: Plavix

SUMMARY:
The aim of this biospecimen repository is to evaluate an individual's genotype, identify the variances, and understand how they relate to treatment with clopidogrel.

DETAILED DESCRIPTION:
The objective of this project is to distinguish genetic profiles that will assist a practitioner in determining the right dose or alternate medication for the patient. In partnership with the genetics team of the Avera Institute for Human Genetics and physicians with the Avera Heart Hospital of South Dakota and North Central Heart Institute, the research team will perform genetic analysis to identify genetic variances.

ELIGIBILITY:
Inclusion Criteria:

* Currently taking or prescribed Clopidogrel or under consideration
* Acute/interventionPatients of the Avera Heart Hospital
* Cardiology clinic patients with the Avera Heart Hospital and North Central Heart Institute

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of either the Avera Heart Hospital of South Dakota or North Central Heart Institute who have been precribed Clopidogrel or are being considered for treatment with Clopidogrel.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gareth Davies, PhD, Principal Investigator — Avera McKennan Hospital & University Health Center
Locations (1):
- Avera Institute for Human Genetics, Sioux Falls, South Dakota, United States

REFERENCES:
- [Background] Topol EJ, Schork NJ. Catapulting clopidogrel pharmacogenomics forward. Nat Med. 2011 Jan;17(1):40-1. doi: 10.1038/nm0111-40. No abstract available. PMID 21217678
- [Background] Mega JL, Hochholzer W, Frelinger AL 3rd, Kluk MJ, Angiolillo DJ, Kereiakes DJ, Isserman S, Rogers WJ, Ruff CT, Contant C, Pencina MJ, Scirica BM, Longtine JA, Michelson AD, Sabatine MS. Dosing clopidogrel based on CYP2C19 genotype and the effect on platelet reactivity in patients with stable cardiovascular disease. JAMA. 2011 Nov 23;306(20):2221-8. doi: 10.1001/jama.2011.1703. Epub 2011 Nov 16. PMID 22088980
- [Background] Shuldiner AR, O'Connell JR, Bliden KP, Gandhi A, Ryan K, Horenstein RB, Damcott CM, Pakyz R, Tantry US, Gibson Q, Pollin TI, Post W, Parsa A, Mitchell BD, Faraday N, Herzog W, Gurbel PA. Association of cytochrome P450 2C19 genotype with the antiplatelet effect and clinical efficacy of clopidogrel therapy. JAMA. 2009 Aug 26;302(8):849-57. doi: 10.1001/jama.2009.1232. PMID 19706858
- [Background] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083
- [Background] Holmes MV, Perel P, Shah T, Hingorani AD, Casas JP. CYP2C19 genotype, clopidogrel metabolism, platelet function, and cardiovascular events: a systematic review and meta-analysis. JAMA. 2011 Dec 28;306(24):2704-14. doi: 10.1001/jama.2011.1880. PMID 22203539